CLINICAL TRIAL: NCT01050894
Title: A Feasibility Study to Determine the Up-regulation of Anti-inflammatory Cytokines in Whole Blood From Patients With Osteoarthritis
Brief Title: Feasibility Study of Anti-inflammatory Cytokines in Whole Blood in Osteoarthritis Patients
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: APS-001
Record Dates: First submitted 2010-01-14; First posted 2010-01-18 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2012-12

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- osteoarthritis patients

SUMMARY:
This is a feasibility study to determine if anti-inflammatory cytokines can be concentrated from patients with osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* radiographic evidence of osteoarthritis
* signed informed consent

Exclusion Criteria:

* Pregnancy
* < 18 years of age
* blood clotting disorder or active hematologic cancer
* undergoing chemotherapy
* history of rheumatoid arthritis
* septic joint or fracture
* active infection or history of chronic infection
* use of cytokine blocking drugs with the last 6 months
* intra-articular steroid or hyaluronic acid (HA) injection within last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with evidence of osteoarthritis.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2010-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Measure anti-inflammatory cytokines | immediately after processing

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - OrthoIndy, Indianapolis, Indiana
  - Orthopaedic Surgery, Kentucky Clinic, Lexington, Kentucky
  - Ohio State University Sports Medicine Center, Columbus, Ohio